CLINICAL TRIAL: NCT00108706
Title: Acute Candesartan Cilexetil Outcomes Stroke Trial (ACCOST)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: City Hospitals Sunderland NHS Foundation Trust (Other)
Collaborators: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACCOST; CTA Number:21763/0001/001; EudraCT Number:2004-001847-31
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Cerebrovascular Accident; Acute Stroke
Keywords: Acute Stroke; Cerebrovascular Accident; Ischaemic Stroke; Candesartan; Angiotensin Receptor Blocker
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — candesartan

INTERVENTIONS:
Drug: Candesartan

SUMMARY:
The aim of this study is to determine whether it is safe and effective to give the Angiotensin Receptor Blocker (ARB) Candesartan within the first 72 hours following acute stroke.

DETAILED DESCRIPTION:
Lowering blood pressure reduces the risk of first ever and recurrent stroke. There is extensive evidence that blood pressure should be lowered following acute stroke, even from so called normal levels. However, it is not clear how soon after acute stroke that blood pressure should be lowered. Observational studies have demonstrated increased mortality with both high and low blood pressure. The optimal management of blood pressure in the immediate post-stroke period remains controversial.

Although uncertainty exists with regard to lowering blood pressure in the acute stages of stroke, two large randomised controlled trials have demonstrated unequivocally that intense management of blood pressure started >4 weeks from the onset of stroke significantly reduces the risk of recurrent stroke. Both of these trials have used an Angiotensin Converting Enzyme Inhibitor (ACE-I) based regime. It has been proposed that these benefits may be due to a direct result of the ACE-I rather than blood pressure lowering per se. Similar vasculoprotective effects have been seen in ARBs, but evidence of their safety and efficacy in acute stroke is limited to those patients with the highest blood pressures (>200/110). The trial (ACCESS) was terminated prematurely due to a positive imbalance in favour of intervention with the ARB Candesartan. If such interventions are to convey potential benefit they need to be started as soon as possible following the acute event in order that the ischaemic cascade which leads to neuronal death may be modified. Further research is first required in order to demonstrate their safety and efficacy when used in this way.

ACCOST is a two phase randomised controlled trial designed to address this important research question. Phase I is a four week double blind placebo controlled phase where patients receive either Candesartan 4 mg daily or matched placebo, with no blood pressure treatment target. A treatment titration step occurs after two weeks where, subject to titration criteria, subjects will receive either Candesartan 8 mg daily or matched placebo. After the first four weeks, the subjects are unblinded and enter Phase II of the trial. Phase II is an eight week open label comparison of Candesartan and 'usual care' with an ACE-I based treatment regime. Blood pressure is now treated to reach the British Hypertension Society target blood pressure of <140/85, with or without additional therapy.

Blinded outcome measures will include neurological recovery based on the National Institutes of Health Stroke Scale, as well as functional recovery. Incidence of first dose hypotension and changes in renal function will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischaemic stroke <72 hours from symptom onset (CT proven)
* Medically stable with no evidence of acute infection and not receiving antibiotic therapy
* Neurologically stable (no progression on NIHSS)
* Able to swallow unthickened fluids safely
* Mean BP (blood pressure) >120/70 in unaffected arm

Exclusion Criteria:

* Previous severe disability (Modified Rankin Score >2)
* Nursing home residents
* Previous history of congestive heart failure requiring treatment with ACE-Inhibitors or angiotensin receptor blockers
* Renal impairment (creatinine >200 mcgmol/L)
* Women of child bearing potential
* Minors <18 years of age
* History of dementia without ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-12; Study Completion 2007-09

PRIMARY OUTCOMES:
Mortality (all causes)
Mortality (vascular causes)

SECONDARY OUTCOMES:
Neurological Recovery (NIHSS [National Institutes of Health Stroke Scale])
Functional Recovery (Modified Rankin/Barthel)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Gray, MD, Principal Investigator — University of Newcastle Upon-Tyne
Locations (1):
- Sunderland Royal Hospital, Sunderland, Tyne and Wear, United Kingdom

REFERENCES:
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Background] PROGRESS Collaborative Group. Randomised trial of a perindopril-based blood-pressure-lowering regimen among 6,105 individuals with previous stroke or transient ischaemic attack. Lancet. 2001 Sep 29;358(9287):1033-41. doi: 10.1016/S0140-6736(01)06178-5. PMID 11589932
- [Background] Schrader J, Luders S, Kulschewski A, Berger J, Zidek W, Treib J, Einhaupl K, Diener HC, Dominiak P; Acute Candesartan Cilexetil Therapy in Stroke Survivors Study Group. The ACCESS Study: evaluation of Acute Candesartan Cilexetil Therapy in Stroke Survivors. Stroke. 2003 Jul;34(7):1699-703. doi: 10.1161/01.STR.0000075777.18006.89. Epub 2003 Jun 19. PMID 12817109